CLINICAL TRIAL: NCT04100265
Title: ANTERO-5: A Clinical Investigation of Gastric Motility in Adult Patients at Risk to Develop Postoperative Ileus Following Colorectal Surgery
Brief Title: ANTERO-5: Gastric Motility in Postoperative Ileus
Acronym: ANTERO-5
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate recruitment due to COVID-19 restrictions.
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: S63029
Record Dates: First submitted 2019-09-11; First posted 2019-09-24 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2019-11

CONDITIONS: Postoperative Ileus

STUDY DESIGN:
Intervention Model Description: Non-randomized investigation in three panels with different eligibility criteria and study procedures.
  The target population in each arm consists of 10 'completers'. Completers are defined as: Panel 1: A successful gastric motility recording of at least 6 hours
  Panel 2: Patients who develop POI (estimated to be 10% of enrolled subjects) and in who gastric motility was recorded successfully for at least 6 hours
  Panel 3: Patients who develop POI, who completed questionnaires for at least 2 days (with a questionnaire completion rate ≥50%).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Panel 1 - High risk for postoperative ileus (Experimental): Intervention in patients at high risk to develop prolonged postoperative ileus. Monitoring postoperative gastric motility for 2 consecutive days in patients who require preventive placement of a nasogastric feeding tube due to a high risk to develop postoperative ileus. Allowing to explore associations between gastric motility and general clinical evolution.
  Interventions: Device: Panel 1 - High risk for postoperative ileus (VIPUN Gastric Monitoring System)
- Panel 2 - Postoperative ileus arm with investigational device (Experimental): Intervention in a population of patients with clinical signs of postoperative ileus, requiring a nasogastric feeding tube for symptom relief. The investigational medical device will be applied. Allowing to explore the association of gastric motility and clinical signs of postoperative ileus in an enriched population with true postoperative ileus.
  Interventions: Device: Panel 2 - Postoperative ileus arm with investigational device (VIPUN Gastric Monitoring System)
- Panel 3 - Postoperative ileus arm with standard of care (No Intervention): Standard of care control group of patients with clinical signs of postoperative ileus requiring a standard nasogastric feeding tube for symptom relief. Symptoms will be surveyed as control group to assess safety and tolerability of the investigational medical device.

INTERVENTIONS:
Device: Panel 1 - High risk for postoperative ileus (VIPUN Gastric Monitoring System) — The VIPUN Gastric Monitoring System prototype 0.3 comprises a nasogastric balloon catheter which is connected to an extracorporeal pressure sensor and data acquisition system. The device is placed during surgery.
  Other Names: VIPUN Gastric Monitoring System prototype 0.3
  Arms: Panel 1 - High risk for postoperative ileus
Device: Panel 2 - Postoperative ileus arm with investigational device (VIPUN Gastric Monitoring System) — The VIPUN Gastric Monitoring System prototype 0.3 comprises a nasogastric balloon catheter which is connected to an extracorporeal pressure sensor and data acquisition system. The device is placed upon the manifestation of clinical signs of postoperative ileus.
  Other Names: VIPUN Gastric Monitoring System prototype 0.3
  Arms: Panel 2 - Postoperative ileus arm with investigational device

SUMMARY:
A monocenter, non-randomized interventional investigation in 3 panels of adult patients undergoing elective colorectal surgery who are at risk to develop postoperative ileus.

The feasibility to use the VIPUN Gastric Monitoring System prototype 0.3 will be explored in this population for the first time.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* At least 18 years old
* BMI between and including 18 and 30
* Understand and able to read Dutch
* Planned to undergo elective colorectal surgery

Exclusion Criteria:

* Known history of documented gastroparesis
* Known history of functional dyspepsia
* Known / suspected current use of illicit drugs
* Known psychiatric or neurological illness
* Any prior gastrointestinal surgery that could influence normal gastric function in the opinion of the investigator
* Known history of heart or vascular diseases like irregular heartbeats, angina or heart attack
* Nasopharyngeal surgery in the last 30 days
* Suspected basal skull fracture or severe maxillofacial trauma
* Known history of thermal or chemical injury to upper respiratory tract or esophagus
* Current esophageal or nasopharyngeal obstruction
* Known coagulopathy
* Known esophageal varices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Feasibility (composite endpoint) | Day 1 - Day 14
  Composite endpoint comprising: procedural success (absence of protocol deviations with regard to motility measurement), tolerability of the device (non-validated questionnaire on nasopharyngeal discomfort and the incidence of intolerance resulting in early removal of the investigational device) and device-related safety (incidence of adverse device effects related to the use of the device).

SECONDARY OUTCOMES:
Gastric motility | Day 1 until termination motility recording (maximum 48 hours)
  Long term motility index
Evolution postoperative ileus - staff reported | Day 1 until completion study procedures (maximum 14 days).
  Incidence of markers of resolution of postoperative ileus (first flatus, bowel sounds, bowel movements, solid food tolerance)
In hospital quality of life (EQ-5D-3L questionnaire) | Day 1 until completion study procedures (maximum 14 days)
  EQ-5D-3L questionnaire consists of 2 pages: EQ-5D descriptive system and an EQ visual analogue scale (EQ VAS).
  EQ-5D-3L (not an acronym) descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The five dimensions can be combined into a 5-digit number that describes the patient's health state. EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'.
Device performance | Day 1 until removal of device, no later than Day 14
  Incidence of device deficiencies
Nausea severity | Day 1 until completion study procedures (maximum 14 days)
  Patient reported severity of nausea (100 mm visual analogue scale ranging from Absent to Worst possible)
Abdominal bloating severity | Day 1 until completion study procedures (maximum 14 days)
  Patient reported severity of abdominal bloating (100 mm visual analogue scale ranging from Absent to Worst possible)
Abdominal pain severity | Day 1 until completion study procedures (maximum 14 days)
  Patient reported severity of abdominal pain (100 mm visual analogue scale ranging from Absent to Worst possible)
Abdominal discomfort severity | Day 1 until completion study procedures (maximum 14 days)
  Patient reported severity of abdominal discomfort (100 mm visual analogue scale ranging from Absent to Worst possible)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No